CLINICAL TRIAL: NCT01905969
Title: Retrospective Validation for Predictive Biomarkers in Stage II/III Gastric Cancer for Adjuvant Chemotherapy With S-1
Brief Title: Predictive Biomarkers in Stage II/III Gastric Cancer for Adjuvant Chemotherapy
Acronym: NJBMR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Iwate Medical University (Other)
Responsible Party: Principal Investigator, Satoshi Nishizuka, Assistant Professor, Iwate Medical University
Other Study IDs: MIAST-NJBMR-12
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Gastric Cancer
Keywords: Gastric caner, adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived paraffin blocks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Biomarker positive: NF-kB(+)/JNK(-) in curatively removed specimens
- Biomarker negative: NF-kB(-)/JNK(+) in curatively removed specimens

SUMMARY:
Adjuvant chemotherapy followed by curative gastrectomy for Stage II/III gastric cancer has improved disease free time and survival. However, there are still considerable number of patients experience relapse even after adjuvant chemotherapy. In an attempt to select patients who really benefit the postoperative adjuvant chemotherapy, we have identified potential biomarkers (NF-kappaB/JNK) from cell line panel screening followed by immunohistochemical validation. In the present study, we further validate the significance of the biomarkers in a larger set of clinical samples to see if chemotherapeutic response can be determined immediately after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed gastric cancer.
* Operated before November 2009.
* Stage Ib/II(except for T1, T3N0)/III.
* Received postoperative (R0) adjuvant chemotherapy (S-1).
* Not received postoperative (R0) adjuvant chemotherapy (surgery alone).
* Signed informed consent to provide paraffin embedded tissue of removed specimens.

Exclusion Criteria:

* With advanced neoplastic lesions other than gastric cancer.
* Paraffin embedded tissue is not available.
* Unknown S-1 treatment condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective study. Data analyses are based on archived record and materials of gastric cancer patients whose treatment was curative surgery followed by adjuvant chemotherapy with S-1.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Iwate Medical University School of Medicine, Morioka, Iwate, Japan

REFERENCES:
- [Background] Ishida K, Nishizuka SS, Chiba T, Ikeda M, Kume K, Endo F, Katagiri H, Matsuo T, Noda H, Iwaya T, Yamada N, Fujiwara H, Takahashi M, Itabashi T, Uesugi N, Maesawa C, Tamura G, Sugai T, Otsuka K, Koeda K, Wakabayashi G. Molecular marker identification for relapse prediction in 5-FU-based adjuvant chemotherapy in gastric and colorectal cancers. PLoS One. 2012;7(8):e43236. doi: 10.1371/journal.pone.0043236. Epub 2012 Aug 14. PMID 22905237